CLINICAL TRIAL: NCT01036009
Title: A Phase II Study of Preemptive Fast Withdrawal of Immunosuppression and Donor Lymphocyte Infusions for Achieving Complete Donor Chimerism Following Allogeneic Transplant for Pediatric Hematologic Malignancies
Brief Title: A Study of Withdrawal of Immunosuppression and Donor Lymphocyte Infusions Following Allogeneic Transplant for Pediatric Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC# 09082; NCT00975598 (obsolete NCT alias)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Acute Leukemia; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Biphenotypic Leukemia; Pre-leukemic Syndromes; Monosomy 7; Bone Marrow Clonal Malformations; Juvenile Myelomonocytic Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia
Keywords: Hematologic; Malignancy; Leukemia; Pre-leukemic; Allogeneic; Transplant; Pediatric
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Chromosome 7, monosomy; Leukemia, Myelomonocytic, Juvenile; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I: Observation (No Intervention): Group I (observation): Patients with full donor chimerism and no evidence of MRD continue to undergo clinical monitoring for acute and chronic graft-vs-host disease and relapse until 3 years post-transplant. Patients undergo repeat chimerism testing at 12 and 24 months post-transplant.
- Group II: Intervention (Experimental): Group II (intervention): Patients undergo withdrawal of immunosuppression and receive donor lymphocyte infusions between days 60-365 post-transplant (or until full donor chimerism is achieved). Patients also undergo clinical monitoring and repeat chimerism testing as in group I.
  Interventions: Other: Withdrawal of immunosuppression and donor lymphocyte infusion

INTERVENTIONS:
Other: Withdrawal of immunosuppression and donor lymphocyte infusion — Intervention will involve fast withdrawal of immunosuppression and DLI until full donor chimerism is achieved.
  Arms: Group II: Intervention

SUMMARY:
There is no curative therapy once acute leukemia patients relapse after transplant. Patients who develop clinically significant graft versus host disease (GVHD) have a lower rate of relapse than those who do not develop GVHD. We are initiating this study of post-transplant fast withdrawal of immunosuppression and donor lymphocyte infusions, with a goal of achieving full donor chimerism in children with hematologic malignancies. If our hypothesis that full donor chimerism results in leukemia-free survival is correct, using immune modulation to achieve full donor chimerism should decrease relapse rate and thus increase survival. The goal of this Phase II study is to identify if achieving full donor chimerism in whole blood CD3+ and leukemia-specific (CD14/15+, CD19+, CD33+ and CD34+) subset may decrease the risk of relapse of patients undergoing allogeneic transplant for hematologic malignancy.

DETAILED DESCRIPTION:
The goal of this Phase II study is to identify if achieving full donor chimerism in whole blood, CD3+, and leukemia-specific subset (CD3+, CD14/15+, CD19+, CD33+ and CD34+ subset) may decrease the risk of relapse of patients undergoing allogeneic transplant for hematologic malignancy.

We estimate that total of 50 recipient patients will need to be enrolled. Of these 50 recipient patients an observation group and an intervention group will be formed. We want to enroll 25 recipient patients in the intervention group, this group will receive study intervention and their outcomes will be the focus of statistical analysis for this study. Intervention will involve fast withdrawal of immunosuppression following transplant and donor lymphocyte infusion (DLI) until full donor chimerism is achieved. Chimerism is a genetic test that measures the proportion of donor's and recipient's cells in blood or bone marrow. Twenty five patients will undergo fast withdrawal of immunosuppression and 33 -50% of them (8-13) will undergo DLI following fast withdrawal of immunosuppression.

Patients will have peripheral blood (PB) chimerism tested upon engraftment. A confirmatory test from PB and bone marrow (BM) will be done on day 45±7. Minimal residual disease (MRD) will be examined by immunoflow, FISH, cytogenetics or PCR. Patients with positive MRD will be on a faster schedule of immune intervention than patients with negative MRD. Interventions will be carried on until 1 year post transplant. If confirmatory testing shows no evidence of MRD and full donor chimerism is present in all subsets, the patient will be part of the "observation" group and be observed until 2 years post transplant. Chimerism will be repeated at 12 and 24 months post transplant. If the patient has mixed chimerism on both confirmatory tests (PB and BM), the patient will be part of the "intervention" group and fast withdrawal of immunosuppression will be initiated. If the patient has mixed chimerism on one of the confirmatory tests (PB or BM), the test will be repeated in 2 weeks and the patient will proceed with either observation or intervention, based on the result of the repeated test. Patients will be followed for the incidence of acute and chronic Graft Versus Host Disease (GVHD) and relapse until 2 years post transplant. The study will be considered successful if the relapse rate at 2 years post transplant is ≤20% for the entire study or ≤ 40% for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months - 25 years.
* Diagnoses of acute leukemia (AML, ALL, biphenotypic leukemia), pre-leukemic syndromes (monosomy 7 or other bone marrow clonal malformations), JMML, myelodysplastic syndromes or CML.
* Undergoing an allogeneic transplant as standard care.
* Performance status: Karnofsky/Lansky>60%.
* Availability of pre-transplant recipient's DNA and donor's DNA for chimerism testing. This could be DNA or material from which DNA could be extracted. Frozen blood would be preferred. For some patients, post transplant specimens that are not infiltrated with donor cells may be used.
* Bone marrow or PBMTC as stem cell source.HLA matching: donor and recipient should be matched at a minimum of 7/8 antigens (A,B,C and DrB1) for bone marrow and PBMTC transplants.
* No history of ≥grade III acute GVHD.

Exclusion Criteria:

* Treatment on other experimental protocols, if withdrawal of immunosuppression interferes with procedures of follow-up on the primary study.
* Leukemia relapse defined as > 5% blasts on bone marrow exam or >1% leukemia cells by immunoflow MRD, or presence of extramedullary leukemia.
* History of acute GVHD ≥ stage III or with any degree of active acute or cGVHD.
* On steroids for any reason.
* Any condition that compromises compliance with the objectives and procedures of this protocol, as judged by the principal investigator.
* Cells for DLI cannot be obtained from the donor.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Horn, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, California
  - All Children's Hospital, St. Petersburg, Florida

REFERENCES:
- [Background] Horn B, Soni S, Khan S, Petrovic A, Breslin N, Cowan M, Pelle-Day G, Cooperstein E, Baxter-Lowe LA. Feasibility study of preemptive withdrawal of immunosuppression based on chimerism testing in children undergoing myeloablative allogeneic transplantation for hematologic malignancies. Bone Marrow Transplant. 2009 Mar;43(6):469-76. doi: 10.1038/bmt.2008.339. Epub 2008 Oct 27. PMID 18955982
- [Derived] Horn B, Petrovic A, Wahlstrom J, Dvorak CC, Kong D, Hwang J, Expose-Spencer J, Gates M, Cowan MJ. Chimerism-based pre-emptive immunotherapy with fast withdrawal of immunosuppression and donor lymphocyte infusions after allogeneic stem cell transplantation for pediatric hematologic malignancies. Biol Blood Marrow Transplant. 2015 Apr;21(4):729-37. doi: 10.1016/j.bbmt.2014.12.029. Epub 2015 Jan 31. PMID 25644958

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 eligible patients relapsed/died before assignment to a study arm
Period: Overall Study
Arm/Group | Group I: Observation | Group II: Intervention
Started | 17 | 26
Completed | 17 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Observation | Group II: Intervention | Total
Number analyzed (Participants) | 17 | 26 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.12 (7.25) | 11.3 (6) | 10.84 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  United States | 17 | 26 | 43

OUTCOME MEASURES:

1. Primary Outcome: Relapse at 2 Years Post-transplant.
Description: Definition of relapse was >5 % blasts in bone marrow
Time Frame: 2 years post transplant.
Measure: Number; unit: participants
Arm/Group | Group I: Observation | Group II: Intervention
Number analyzed (Participants) | 17 | 26
participants | 6 | 4

2. Secondary Outcome: 2 Years Post-transplant Survival.
Time Frame: 2 years post transplant
Measure: Number; unit: participants
Arm/Group | Group I: Observation | Group II: Intervention
Number analyzed (Participants) | 17 | 26
participants | 11 | 21

3. Secondary Outcome: The Incidence of Acute Graft Versus Host Disease (aGVHD).
Description: Definition and diagnostic criteria of aGVHD according to: 1994 Consensus Conference on Acute GVHD Grading. Przepiorka D1, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. Bone Marrow Transplant. 1995 Jun;15(6):825-8.
  In this system, patients are divided into one of four grades (I-IV) depending on the degree, or stage, of involvement in three organs. The skin is staged with percent body surface involved, the liver is staged with degree of bilirubin elevation, and the gastrointestinal tract is staged with amount of diarrhea.
Time Frame: 2 years post transplant
Measure: Number; unit: participants
Arm/Group | Group I: Observation | Group II: Intervention
Number analyzed (Participants) | 17 | 26
participants | 11 | 5

4. Secondary Outcome: The Incidence of Chronic GVHD (cGVHD).
Description: Diagnostic criteria of cGVHD from: Filipovich AH, Weisdorf D, Pavletic S et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-host disease: I Diagnosis and Staging Working Group Report. Biology of Blood and Marrow Transplantation 2005;11:945-955.
  The diagnosis of chronic GVHD requires the following:
  1) Distinction from acute GVHD; 2) Presence of at least 1 diagnostic clinical sign of chronic GVHD or presence of at least 1 distinctive manifestation confirmed by pertinent biopsy or other relevant tests; 3) Exclusion of other possible diagnoses.
  Scoring of organ manifestations requires careful assessment of signs, symptoms, laboratory values, and other study results. A clinical scoring system (0-3) is used for evaluation of the involvement of individual organs and sites. Global assessment of severity (mild, moderate, or severe) is derived by combining organ- and site-specific scores.
Time Frame: 2 years post transplant
Measure: Number; unit: participants
Arm/Group | Group I: Observation | Group II: Intervention
Number analyzed (Participants) | 17 | 26
participants | 6 | 2

5. Post Hoc Outcome: Late Relapses
Description: The number of patients who relapsed after 2-year primary endpoint. To assess a potential for late relapse-rate in the intervention arm only, patients in the intervention arm were provided additional follow-up until 3-yrs post transplant. The criterion for relapse was >5% blasts in bone marrow.
Time Frame: 24-36 months post-transplant
Population: surviving patients in the intervention arm who had not relapsed as of 24 months were followed for an additional 12 months (until 3 years post-transplant)
Measure: Number; unit: participants
Arm/Group | Group II: Intervention
Number analyzed (Participants) | 21
participants | 4

6. Post Hoc Outcome: Time Until Late Relapse
Description: Number of months post-transplant until late relapse, in intervention patients relapsing after the 2-year primary study endpoint. Relapse defined as >5% blasts in bone marrow
Time Frame: 24-36 months post-transplant
Population: intervention patients who relapsed after the 2 year primary study endpoint
Measure: Mean (Full Range); unit: months
Arm/Group | Group II: Intervention
Number analyzed (Participants) | 4
months | 32.025 [25 to 36.32]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Due to the severity of illness in this patient population, this study collected and reported Adverse Events only if at least possibly related to study participation, and only in patients undergoing study intervention (intervention arm).
Arm/Group | Group I: Observation | Group II: Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/26
Other Adverse Events (participants affected / at risk) | 0/0 | 9/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I: Observation (N=0) | Group II: Intervention (N=26)
intervention-related-death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — severe cGVHD that involved lungs, treated with Prednisone, death due to fungal lung infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I: Observation (N=0) | Group II: Intervention (N=26)
aGVHD grade I-III (Immune system disorders) | 0 (0) | 3 (3)
cGVHD (Immune system disorders) | 0 (0) | 2 (2)
progressive disease (Blood and lymphatic system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes